CLINICAL TRIAL: NCT04898465
Title: Improving Family's Adherence to Dental Care After Dental General Anaesthesia (DGA). Helsinki Early Childhood Caries - Child Abuse and Neglect-study. (HECC-CAN)
Brief Title: Improving Family's Adherence to Dental Care After DGA (HECC-CAN-study)
Acronym: HECC-CAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Heikki Alapulli, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HUS/180/220
Record Dates: First submitted 2021-05-03; First posted 2021-05-24 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Dental Caries; Child Neglect
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social Paediatric Intervention (Experimental): Multiprofessional social paediatric meeting with the family.
  Interventions: Other: Social Paediatric Intervention
- Control group (No Intervention): Normal post-DGA dental programme.

INTERVENTIONS:
Other: Social Paediatric Intervention — Family will meet the hospital's social-paediatrician and social worker. Together they will evaluate the need for social support, risk for neglect and refer families for local social services if needed. The visit will contain primary and secondary prophylaxis of child abuse and neglect.
  Arms: Social Paediatric Intervention

SUMMARY:
Early childhood caries (ECC) is a common disease. Its prevalence is highest in poor, socially disadvantaged, and minority groups. Dental treatment under General Anaesthesia (DGA) is common, especially among the youngest patients. Parental adherence to child's post-DGA dental treatment is varying. Non-attendance to preventive care appointments and dental check-ups after the DGA is also common. The primary aim of this study is to explore if a multi-professional (paediatrician and social worker) intervention after the child's DGA can increase the adherence to post-DGA dental care. The secondary aim is to compare its possible influence on children's oral health 18 months after the DGA. Our hypothesis is that multi-professional counselling and support after the DGA will lead to better adherence to the scheduled preventive dental programme and better oral health for these children in the long run.

DETAILED DESCRIPTION:
In an earlier Finnish study 26% of the children did not attend to their first scheduled appointment after the DGA and during a four years follow-up period 63% of the patients had one or more no-shows.

Based on the assumption that reducing the amount of no-shows to half of the reported earlier (60% vs. 30%) is a clinically relevant result, we need 42 patients for both groups (alpha 0.05, beta 0.2, power 0.8).

ELIGIBILITY:
Inclusion Criteria:

* reason for DGA is dental caries
* place of birth is Finland
* primary dentition

Exclusion Criteria:

* chronic disease which needs treatment in tertiary hospital

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Number of uncancelled dental appointments after DGA | 0-18 months after the DGA
  Amount of unused or uncancelled dental appointment times after DGA

SECONDARY OUTCOMES:
Number of new decayed teeth after DGA | 0-18 months after the DGA
  Amount of caries lesions observed after DGA

CONTACTS AND LOCATIONS:
Overall Officials: Eeva Nikkola, MD, PhD, Principal Investigator — Consultant
Locations (1):
- New Children's Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Savanheimo N, Vehkalahti MM. Five-year follow-up of children receiving comprehensive dental care under general anesthesia. BMC Oral Health. 2014 Dec 15;14:154. doi: 10.1186/1472-6831-14-154. PMID 25512015